CLINICAL TRIAL: NCT01543945
Title: Prevention Post Operative Nausea Vomiting in Ambulatory Gynecologic Laparoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Thanyamon Asampinwat, Assistant Professor, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PONV9268
Record Dates: First submitted 2012-02-28; First posted 2012-03-05 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: Postoperative Nausea and Vomiting; Ambulatory; Gynecologic laparoscopy; Incidence of postoperative nausea and vomiting.
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Vomiting | interventions — Dexamethasone; Ondansetron; Dimenhydrinate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multimodal antiemetic management group (Experimental): Multimodal antiemetic group : Low risk :no PONV prophylaxis moderate risk : ondansetron 4 mg iv high risk : dexamethasone 4 mg + ondansetron 4 mg Extremely high risk : dexamethasone 4 mg + ondansetron 4 mg + dimenhydrinate 1 mg
  Interventions: Drug: Dexamethasone; Drug: Ondansetron; Drug: Dimenhydrinate
- Control group (Active Comparator): Control group: Low and moderate risk : no PONV prophylaxis High risk : Ondansetron 4 mg. iv Extremely high risk : Ondansetron 4 mg .iv
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Dexamethasone — 4 mg iv before induction for high and extremely high risk
  Other Names: Multimodal antiemetic group :; high risk : dexamethasone 4 mg + ondansetron 4 mg; Extremely high risk : dexamethasone 4 mg +; ondansetron 4 mg +; dimenhydrinate 1 mg
  Arms: Multimodal antiemetic management group
Drug: Ondansetron — 4 mg iv before ended surgery 30 min
Drug: Dimenhydrinate — 1 mg/kg iv before ended surgery 30 min
  Arms: Multimodal antiemetic management group

SUMMARY:
The purpose of this study is to compare the incidence of Postoperative nausea and vomiting between the intervention group who received multimodal antiemetic management and the control group who did not get this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory gynecologic laparoscopy
* Age 18-45 years
* ASA class 1-2

Exclusion Criteria:

* The patients who take opioid, steroid, pyschotics or antiemetic drug within 24 hours before surgery
* History of antiemetic, anesthetic and analgesic drugs allergy
* Pregnancy or breast feeding
* Body mass index >34 kg/square metre

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 340 (Actual)
Dates: Start 2008-03; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Incidence of PONV in ambulatory gynecologic laparoscopy | four year

CONTACTS AND LOCATIONS:
Overall Officials: Thanyamon Asampinwat, MD, Principal Investigator — Anesthesiology department, Faculty of Medicine, Prince of Songkla University Thailand
Locations (1):
- Anesthesiology Department, Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand